CLINICAL TRIAL: NCT03565029
Title: Total Neoadjuvant Treatment Without Surgery For Locally Advanced Rectal Cancer: Prospective Clinical Trial To Assess Tumor Complete Response, Circulating Tumor Genetic And Epigenetic Biomarkers, And Stromal Transcriptome To Interpret Clinical Outcome
Brief Title: Total Neoadjuvant Treatment Without Surgery For Locally Advanced Rectal Cancer
Acronym: NO-CUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003671-60
Record Dates: First submitted 2018-06-08; First posted 2018-06-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Colo-rectal Cancer
Keywords: rectal cancer; neoadjuvant; non operative management
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — XELOX; Radiotherapy

STUDY DESIGN:
Intervention Model Description: one-stage phase II trial seeking to establish whether an oxaliplatin-based chemotherapy preceding standard neo-adjuvant fluoropyrimidines-based chemo radiotherapy, can safely spare demolitive surgical intervention in patients with operable rectal cancer, without increasing the risk of distant relapse. The trial also has a translational component aimed at establishing whether selected genomic, epigenetic, and transcriptomic markers are predictive of tumor and patient outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Medium/low locally advanced rectal cancer (Experimental): Patients with Stage II (cT3-4 N0) or Stage III (cT1-4, N1-3) locally advanced rectal cancer amenable to Total Mesorectal Excision (TME)/Abdominal-Perineal Amputation
  Interventions: Drug: XELOX; Radiation: Radiotherapy

INTERVENTIONS:
Drug: XELOX — Capecitabine and Oxaliplatin (4x cycles)
Radiation: Radiotherapy — Pelvic radiotherapy

SUMMARY:
NO-CUT is a one-stage phase II trial seeking to establish whether an oxaliplatin-based chemotherapy preceding standard neo-adjuvant fluoropyrimidines-based chemo radiotherapy, can safely spare demolitive surgical intervention in patients with operable rectal cancer, without increasing the risk of distant relapse. The trial also has a translational component aimed at establishing whether selected genomic, epigenetic, and transcriptomic markers are predictive of tumor and patient outcome.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer worldwide and the second leading cause of cancer death in Europe. Rectal cancer accounts for about 25-30% of all colorectal cancer diagnoses. Five-year survival rates depend on stage at diagnosis, about 92% for stage I, 87% for stage II A, 63% for stage II B, 89% for stage III A, 69% for stage III B, and for stage III C cancers the survival rate is about 53%; stage IV rectal cancers have a 5-year relative survival rate of about 11%. With the chemoradiation therapy (CRT), the resulting pathologic complete response (pCR) across all stages has been documented in up to 30% of patients. Most importantly, patients achieving pCR have lower rates of tumor recurrence, and improved survival, compared to those who do not achieve pCR. Moreover, data from the National Surgical Quality Improvement Project document a 35% risk of morbidity associated with both low anterior and abdominoperineal resection. Long-term morbidity includes bowel and bladder incontinence, sexual dysfunction, and complications associated with temporary and permanent stomas.

Due to the observation of the absence of residual tumor in the pathological specimens of a significant proportion of patients treated with CRT for local or locally advanced rectal cancer, in the early-2000s, two clinical issues arose: firstly, if pCR could be predicted after CRT with clinical, radiological, or endoscopic restaging assessment thus defining clinical complete response (cCR); and secondly if patients with cCR should necessarily undergo radical surgery to achieve cure at the cost of morbidity, mortality, and functional consequences associated with radical rectal surgery. Consequently, an increasing number of reports suggested that non-operative management (NOM), consisting of close surveillance of patients with cCR, could be an acceptable alternative to rectal surgery (proctectomy). Led by small prospective series published since the late 90's by Habr-Gama and colleagues, several small international series have reported similar oncologic outcomes in cCR patients followed by close active surveillance (the so-called watch-and-wait (W&W) or NOM approach) compared to those treated with radical surgery.

Between 2011 and 2013 a NOM approach was carried out in 31 patients achieving cCR out of 259 (12%). In their analysis, a further 98 patients, selected from a United Kingdom regional registry, similarly managed from 2005 to 2015, were added to the NOM group (129 patients). Overall Survival and Disease Free Survival rates resulted at least comparable to that of patients treated with standard surgery following neo-adjuvant CRT.

On the other hand, these small single institution pilot studies have been conducted enrolling small cohorts of patients with less than 500 patients having been evaluated worldwide. A high variability in stage at diagnoses, local recurrence rate, distant recurrence rate (0-60% and 0-17%, respectively) and type and outcome of salvage therapy (0 to 100%) have been reported and no reliable data on long term outcomes are available. Based on these limitations, the NOM of rectal cancer deserves consideration within purposely designed clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the medium/lower rectum
* Patients must have Stage II (cT3-4 N0) or Stage III (cT1-4, N1-3) tumor
* Locally advanced rectal cancer amenable to Total Mesorectal Excision (TME)/Abdominal-Perineal Amputation
* No evidence of distant metastases by chest, abdomen, and pelvis contrast enhanced CT scan (TC-positron emission computed tomography (PET) Whole Body (WB) is acceptable alternative in patient allergic to iodate contrast medium)
* No prior pelvic radiation therapy
* No prior oncologic medical therapy or surgery for rectal cancer
* Age >18 years
* No infections requiring systemic antibiotic treatment
* Performance status 0-1 (ECOG Scale)
* absolute neutrophil count (ANC) > 1.5 cell/mm3, Hb>8.0 g/ dL, Platelet Count (PLT)>150,000/mm3, total bilirubin < or equal or 1.5 x upper limit of normal, Aspartate Aminotransferase (AST) < or equal to three times upper limit of normal, Alanine Aminotransferase (ALT)< or equal to three times upper limit of normal; Serum creatinine level < or equal to 1.5 times the upper limit of normal
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation
* Women with childbearing potential who are negative for pregnancy test (urine or blood) and who agree to use effective contraceptive methods
* Male subjects must also agree to use effective contraception

Exclusion Criteria:

* Recurrent rectal cancer
* Patients with a history of any arterial thrombotic event within the past 6 months, including angina (stable or unstable), MI, or CVA
* Intolerance or contraindication to Magnetic Resonance (MR) procedure
* Patients with any other concurrent medical or psychiatric condition
* Gastro-intestinal abnormalities, inability to take oral medication, any condition affecting absorption
* Patients with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer.
* Patients with a history of thrombotic episodes, such as deep venous thrombosis, pulmonary embolus, Myocardial Infarction (MI) or cerebral vascular accident (CVA) occurring more than 6 months prior to enrollment may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Patients who are anticoagulated for atrial fibrillation or other conditions may participate, provided they are on stable doses of anticoagulant therapy.
* Patients receiving other anticancer or experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Distant Relapse-Free Survival (DRFS) | 2.5 years
  Disease free survival rate

SECONDARY OUTCOMES:
Clinical complete response rate | 2 months
  Clinical complete response rate
Local recurrence and organ preservation rate | 6 months
  Local recurrence and organ preservation rate
Colostomy-free survival | 6 months
  Colostomy-free survival
Overall survival | 2.5 years
  Overall survival
Patient reported outcomes | 2.5 years
  European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire-C30 and its colorectal cancer specific module Quality of Life Questionnaire-38)

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Weekly Scientific Board Commission meetings
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Weekly